CLINICAL TRIAL: NCT00671580
Title: A Phase II Randomized, Observer-Blind, Multi-Center Study to Evaluate the Safety, Potential Efficacy, and Pharmacokinetics of Two Dosing Regimens of Intravenous PZ-601 and Standard of Care in the Treatment of Complicated Skin and Skin Structure Infections
Brief Title: Safety, Potential Efficacy, and Pharmacokinetics of PZ-601 in the Treatment of Complicated Skin and Skin Structure Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Protez Pharmaceuticals, Inc. (Industry)
Responsible Party: Shelley Fayocavitz, Associate Director, Clinical Study Management, Protez Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PZ-601-02
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Skin Infections
Keywords: Skin Infections; Complicated Skin and Skin Structure Infections
MeSH Terms: conditions — Cellulitis | interventions — SM-216601; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): PZ-601
  Interventions: Drug: PZ-601
- B (Experimental): PZ-601
  Interventions: Drug: PZ-601
- C (Active Comparator): Standard of Care
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: PZ-601 — 750 mg
  Arms: A
Drug: PZ-601 — 1000 mg
  Arms: B
Drug: Standard of Care — as directed
  Arms: C

SUMMARY:
The purpose of this study is to evaluate the potential effect and safety of two different doses of PZ-601 and to compare this with another antibiotic that is approved by the US Food and Drug Administration (also known as FDA) to treat adults with skin and skin structure infections.

DETAILED DESCRIPTION:
PZ-601 is a novel investigational carbapenem antibiotic with an antimicrobial spectrum of activity that includes pathogens responsible for community-acquired bacterial infections as well as multidrug-resistant Gram-positive pathogens - MRSA and vancomycin-resistant enterococci. PZ-601 also has activity against Gram-negative organisms including cephalosporin and quinolone resistant Enterobacteriaceae as well as Bacteriodes fragilis and peptostreptococci. Based on the antimicrobial profile, PZ-601 is a potentially promising agent for the treatment of complicated skin and skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided by the patient
2. Males and females ≥ 18 years of age
3. Diagnosis of complicated skin and skin structure infection defined as infection which meets the following criteria:

   * Suspected to be caused by bacterial pathogens, including multi-drug resistant organisms such as MRSA, and
   * Involves deeper soft tissue and/or require significant surgical intervention such as:

     * major abscesses
     * infected burn (less than or equal to 20% body surface area)
     * traumatic wound infection
     * deep/extensive cellulitis
     * surgical wound infection
     * infected ulcer (with the exception of multiple infected ulcers at distant sites.) Please Note: Patients with multiple sites of skin infection may be enrolled in the study. The most severely affected site or the one most likely to yield a positive culture should be chosen to follow throughout the course of evaluations.
4. Presents with at least TWO of the following local symptoms:

   * Purulent or seropurulent drainage/discharge
   * Erythema
   * Fluctuance
   * Heat/Localized Warmth
   * Pain/tenderness to palpation
   * Swelling/induration
5. At least ONE of the following systemic signs of infection

   * Increased Temperature (≥100.4ºF/≥38.0ºC) measured orally or its equivalent (note: other methods of obtaining temperature are acceptable)
   * WBC (>10,000 cells/mm3)
   * Immature neutrophils (>10% band forms regardless of the total peripheral white count)
6. Require initial hospitalization with at least 7 days of parenteral therapy for treatment of suspected cSSSI infection
7. Ability to obtain a culture and Gram stain of the cSSSI site within 48 hours prior to the initiation of study medication;

Exclusion Criteria:

1. Female patients who are pregnant, lactating (breast milk feeding), or planning a pregnancy during the course of the study, or who are of child bearing potential and not using an acceptable method of birth control (ie, surgically sterile, intrauterine device, oral contraceptive plus barrier contraceptive, hormone delivery system plus barrier contraceptive or condom in combination with contraceptive cream, jelly or foam)
2. Received more than 24 hours of systemic antibiotic therapy within 96 hours of initiation of study medication for the current episode of cSSSI, unless:

   * there is evidence of clinical failure following at least 48 hours of prior, non-study systemic therapy OR
   * there is microbiological evidence of failure (ie, Gram stain reveals WBC and at least one potential pathogen or isolation of an organism resistant to the prior therapy)
3. Concomitant conditions requiring antimicrobial therapy that would interfere with the evaluability of the condition under study
4. Anticipated need for prolonged antibiotic therapy (ie, >14 days)
5. Topical use of antimicrobials (excluding vaginally or topically administered antifungal agents)
6. cSSSI known or suspected to be caused by fungal, parasitic or viral infections
7. cSSSI of the following categories:

   * infected diabetic foot ulcers or decubitus ulcer
   * multiple infected ulcers at distant sites
   * involve an ischemic ulcer due to peripheral vascular disease
   * presence of gangrene of any etiology
8. Necrotizing fasciitis or gas gangrene
9. Infections resulting from human or animal bites (excluding infections secondary to arthropod bites)
10. Known or suspected osteomyelitis or septic arthritis
11. Superinfected eczema or other chronic medical conditions (eg, atopic dermatitis, hidradentitis suppurativa) characterized by prominent signs of inflammation for an extended period even after successful bacterial eradication
12. Patients who have undergone more than two surgical interventions (defined as surgery that cannot be performed at the bedside) for treatment of cSSSI at the time of enrollment
13. Patients who are expected to require more than two surgical interventions (defined as surgery that cannot be performed at the bedside) for treatment of cSSSI during the first 48 hours following study enrollment
14. Infections complicated by the presence of prosthetic materials that will not be removed such as permanent intracardiac devices or joint replacement prosthesis
15. Moderately or severely impaired renal function with known creatinine clearance <50 mL/min (based on the Cockcroft-Gault formula using ideal body weight)
16. ALT or AST >3x upper limit of normal or bilirubin >1.5x upper limit of normal (ULN)
17. Neutropenia defined as an absolute neutrophil count <500/mm3
18. Thrombocytopenia defined as a platelet count <50,000 cells/mm3
19. Infection with human immunodeficiency virus and a CD4 count known at the time of enrollment to be <200 cells/mm3 or another Acquired Immune Deficiency Syndrome (AIDS)-defining illness
20. Requiring concomitant administration of systemic corticosteroids greater than 40 mg/day of prednisolone (or equivalent)
21. Treatment with cancer chemotherapy, radiotherapy, or potent, non-corticosteroid immunosuppressant drugs (eg, cyclosporine, azathioprine, tacrolimus, immune-modulating monoclonal antibody therapy, etc.) within the 3 months prior to study enrollment
22. Concomitant therapy with medications known to lower seizure threshold or those patients with a history of seizure disorder
23. Concomitant therapy with medications known to be associated with QTc prolongation potential (eg, Class IA and Class III anti-arrhythmic agents)
24. History or significant cardiac disease defined by the following:

    * New York Heart Association (NYHA) Class III or IV heart failure
    * History or risk of ventricular arrhythmia (excluding isolated premature ventricular contractions [PVC's] or consecutive PVC's <10 beats), Torsades de Pointes, 2nd or 3rd degree AV block, or QTc interval >470 mm/sec
25. History of any hypersensitivity or allergic reaction to beta-lactam drugs such as carbapenems, penicillins, or cephalosporins
26. History of any hypersensitivity or allergic reaction to vancomycin or history of Red Man Syndrome
27. Any planned medical intervention or personal event that might interfere with the ability to comply with the study requirements
28. Any condition that, in the opinion of the principal investigator, would compromise the safety of the patient or the quality of the data
29. Life expectancy of less than 3 months from the time of enrollment
30. Use of an investigational drug or device (ie, a drug or device without an FDA approved indication) within the previous 30 days
31. Prior participation in this protocol
32. Unable or unwilling to adhere to the study-specified procedures and restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter is the proportion of patients experiencing clinical response based on improvement or resolution of clinical signs and symptoms of infection in the Clinically Evaluable population at the Test of Cure visit. | up to 6 weeks

SECONDARY OUTCOMES:
Clinical Response in the Clinically Evaluable (CE) population at the End of Treatment (EOT) visit | Up to 4 weeks
Clinical Response in the Intent-to-Treat (ITT), Microbiological ITT (mITT), and Microbiologically Evaluable (ME) populations at the Test of Cure (TOC) visit | Up to 4 weeks
Clinical Response in the Intent-to-Treat (ITT), Microbiological ITT (mITT), and Microbiologically Evaluable (ME) populations at the End of Treatment (EOT) visit | Up to 4 weeks
By-pathogen and by-patient Microbiological Response in the Microbiological ITT (mITT) and Microbiologically Evaluable (ME) populations at the Test of Cure (TOC) visit | Up to 4 weeks
By-pathogen and by-patient Microbiological Response in the Microbiological ITT (mITT) and Microbiologically Evaluable (ME) populations at the End of Treatment (EOT) visit | Up to 4 weeks
Overall combined Clinical and Microbiological Response in the Microbiological ITT (mITT) and Microbiologically Evaluable (ME) populations at the Test of Cure (TOC) visit | Up to 4 weeks
Overall combined Clinical and Microbiological Response in the Microbiological ITT (mITT) and Microbiologically Evaluable (ME) populations at the End of Therapy (EOT) visit | Up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - eStudySite - Sharp Chula Vista, Chula Vista, California
  - Novellus Research Site, Fountain Valley, California
  - Novellus Research Site, Long Beach, California
  - eStudySite - Tri-City Medical Center, Oceanside, California
  - eStudySite - Good Samaritan Hospital, San Jose, California
  - Infectious Disease of Indiana, PSC, Indianapolis, Indiana
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - University of Missouri Health Care, Columbia, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Holy Name Hospital Institute for Clinical Research, Teaneck, New Jersey
  - Summa Health System, Akron, Ohio
  - Remington-Davis, Inc., Columbus, Ohio
  - NewBridge Medical Research, Warren, Pennsylvania